CLINICAL TRIAL: NCT02663076
Title: Factor XA - Inhibition in RENal Patients With Non-valvular Atrial Fibrillation - Observational Registry
Acronym: XARENO
Status: Completed | Type: Observational
Sponsor: GWT-TUD GmbH (Other)
Collaborators: ClinStat GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: XARENO-Registry
Record Dates: First submitted 2015-12-17; First posted 2016-01-26 (Estimated); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- VKA - Vitamin K antagonist group: VKAs used in correspondence with the national guidelines for therapy of NVAF in the respective country.
- Rivaroxaban group: Rivaroxaban used in correspondence with the national guidelines for therapy of NVAF in the respective country.
- noAC group: noAC used in correspondence with the national guidelines for therapy of NVAF in the respective country.

SUMMARY:
The multicenter registry will collect clinical data from 1600 patients with non valvular atrial fibrillation (NVAF) and chronic kidney disease (eGFR 15-49 mL/min per 1.73 m2).

The overall objective of this registry is to assess chronic kidney disease (CKD) progression and clinical outcomes with regard to anticoagulation strategies in NVAF patients with eGFR 15-49 mL/min per 1.73 m2 in routine clinical practice.

DETAILED DESCRIPTION:
This is a prospective registry allowing a structured, non-interventional collection of data. Participating physicians will not be subject to any instructions with regard to the diagnosis and therapy of their patients. All patient treatment is carried out within clinical routine, at the discretion of the physician and according to existing treatment guidelines.

This registry will be carried out as an investigator-initiated, multicentre, prospective, non-interventional and observational registry at approximately 160 sites in Germany, Austria, Switzerland, France, Belgium and Luxembourg.

The registry will collect clinical data of approximately 1600 patients with CKD (eGFR 15-49 mL/min per 1.73 m2) and NVAF receiving rivaroxaban, OAC with VKA, or no AC therapy, who are prospectively followed for a flexible duration with a minimal follow-up duration of 12 months until study end is announced (planned minimum 360 days / planned maximum 84 months).

The plan of the registry is to include at least 1600 patients with CKD and NVAF and rivaroxaban therapy or VKA therapy or no AC therapy.

The aim is to include at least 700 patients with rivaroxaban therapy and VKA therapy, respectively. Into the exploratory treatment arm of patients receiving no AC therapy about 100 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients, age ≥ 18 years
* CKD with eGFR 15 - 49 mL/min per 1.73 m2
* non-valvular atrial fibrillation (NVAF) with indication for anticoagulation therapy
* a treatment strategy for the ≥ 3 previous months before enrolment with either: rivaroxaban or VKA (OAC cohorts) or no anticoagulation (no AC cohort)
* informed consent
* availability for follow up
* life expectancy of ≥6 months

Exclusion Criteria:

* exclusion criteria according to the local product information for the respective anticoagulation treatment
* planned treatment with other anticoagulants
* expected renal-replacement therapy within the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CKD (eGFR15-49 mL/min per 1.73 m2) and NVAF are in the focus of the XARENO registry
Sampling Method: Probability Sample
Enrollment: 1700 (Actual)
Dates: Start 2016-04; Primary Completion 2022-01 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
decline in eGFR in mL/min per 1.73 m2 | 12 month
major bleeding | 12 month
all-cause mortality | 12 month
TIA, stroke or systemic arterial embolism | 12 month
major cardiovascular events (MACE) | 12 month
symptomatic venous thromboembolic events | 12 month
net-clinical benefit (stroke and other thromboembolic events, major bleeding, and all-cause mortality) | 12 month

SECONDARY OUTCOMES:
initiation of chronic renal replacement therapy | 12 month
eGFR < 15 mL/min per 1.73 m2 (CKD Stage 5 Dialysis and Non-Dialysis) | 12 month
eGFR decline of ≥ 30% | 12 month
doubling of serum creatine concentration | 12 month
acute kidney injury (AKI) events defined as acute kidney injury associated with either hospitalization or emergency department visit, where AKI event is the lead diagnosis | 12 month, 18 month
rates of hospitalizations | 12 month, 18 month
length of hospitalizations | 12 month, 18 month
causes of hospitalizations | 12 month, 18 month
persistence with OAC therapy | 12 month, 18 month
reasons for OAC therapy discontinuation | 12 month, 18 month
  descriptive analysis of reasons for therapy discontinuation (verbal description by investigator)

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Kreutz, Prof. Dr., Study Director — Charite University, Berlin, Germany; Jan Beyer-Westendorf, PD Dr., Study Chair — University Clinic Technical University Dresden
Locations (118):
- Austria (8):
  - Krankenhaus St. Josef Braunau, Braunau am Inn
  - Medizinische Universitätsklinik, Graz
  - Allgemeines Krankenhaus der STadt Linz, Linz
  - Krankenhaus der Elisabethinen Linz, Linz
  - Medizinische Universität Wien, Vienna
  - Meidzinische Universität Wien, Vienna
  - Sozialmedizinischer Zentrum-Süd Kaiser-Franz-Josef-Spital, Vienna
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhügel, Vienna
- Belgium (7):
  - Centre Hospitalier EpiCURA-Baudour, Baudour
  - CUB Hôpital ERASME, Brussels
  - CHU de Charleroi, Charleroi
  - Centre Hospitalier Régional de la Citadelle, Liège
  - Centre Hospitalier Chrétien (CHC) St Joseph, Liège
  - Centre Hospitalier Universiatire du SART-TILMAN, Liège
  - Centre Hospitalier de Wallonie Picarde (Chwapi), Tournai
- France (26):
  - Clinique Sainte-Isabelle, Abbeville
  - CH Abbeville, Abbeville
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CH Argenteuil Centre Hospitalier Victor Dupouy, Argenteuil
  - CHU Avicenne (AP-HP), Bobigny
  - CHU Bordeaux-Hôpital Saint André, Bordeaux
  - CHU Bordeaux-Hôpital Pellegrin, Bordeaux
  - CHRU Brest-Hôpital la Cavale Blanche, Brest
  - CH Cholet, Cholet
  - CHU Clermont Ferrand, Clermont-Ferrand
  - Hôpital Louis Mourier (AP-HP), Colombes
  - CH de Compiègne-Noyon (CHNC), Compiègne
  - Hôpital Henri Mondor (AP-HP), Créteil
  - CHD Vendée, La Roche-sur-Yon
  - CHG de Chartres-Hôpital Général Louis Pasteur, Le Coudray
  - CHR Metz-Thionville, Hôpital de Mercy, Metz
  - CHU Nantes-site Hotel Dieu, Nantes
  - CHU Carémeau, Nîmes
  - Pitié-Salpètrière Hospital (AP-HP), Paris
  - Claude Bernard - Bichat Hospital, Paris
  - Hôpital Bretonneau (AP-HP), Paris
  - CHU Nantes-Hôpital nord Laennec, Saint-Herblain
  - CHRU Strasbourg Nouvel Hôpital Civil, Strasbourg
  - CHI Toulon La Seyne sur mer - Hopital Sainte Musse, Toulon
  - Hôpital Nord Franche Comté, Trévenans
- Germany (74):
  - Kardiologische Praxis, Bad Homburg
  - Schilddrüsenzentrum Bergstrasse/Praxis Innere Medizin, Bensheim
  - FA für Innere Medizin, Bergisch Gladbach
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Franziskus-Krankenhaus Berlin, Berlin
  - Praxis Rankestrasse, Berlin
  - MVZ Dres. Ramdohr, Berlin
  - St. Joseph Krankenhaus Berlin-Tempelhof GmbH, Berlin
  - Facharzt für Allgemeinmedizin, Berlin
  - Praxis, Berlin
  - Kardiologische Arztpraxis, Borsdorf
  - Studienzentrum Schwittay, Böhlen
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Krankenhaus Buchholz, Buchholz
  - Gemeinschaftspraxis Kellner und Ehrhardt, Camburg
  - Klinikum Coburg GmbH, Coburg
  - Uniklinik Köln, Cologne
  - Kardiologische Partnerschaftsgesellschaft, Cottbus
  - ZID- Zentrum für Innere Medizin Dachau, Dachau
  - Kardiovaskuläres Zentrum Darmstadt, Darmstadt
  - Klinikum Dortmund GmbH, Dortmund
  - Kardiologie Dortmund, Dortmund
  - Nephrologische Praxis, Dortmund
  - Praxisklinik Herzkreislauf am Wasaplatz, Dresden
  - Praxis Dr. med Steffen Fischer, Dresden
  - Praxis Dr. med. Christoph Axthelm & Kollegen, Dresden
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Gemeinschaftspraxis Dr. med. Sybille Jänsch, Dresden
  - Praxis Dr. med. Frank Richard, Erfurt
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Gemeinschaftspraxis im Altstadtcarree, Kardiologie, Fulda
  - MVZ Prof. Mathey, Prof. Schofer GmbH, Hamburg
  - Herzpraxis Altona, Hamburg
  - Zentrum für Nieren-, Hochdruck und Stoffwechselerkrankungen, Hanover
  - DOKUSAN, Herne
  - Universitätsklinikum des Saarlandes, Homburg
  - Praxisnetz Dr. Haaß & Kollegen, Inden
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Studienzentrum Dr. med. Karl-Friedrich Appel, Kassel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Gemeinschaftspraxis Wittwer, Bargemann, Baar, Kiel
  - Gemeinschaftspraxis Scheuermann & Persicke, Kornwestheim
  - Praxis, Königsbrück
  - Eickenhof Dialyse - Gemeinschaftspraxis, Langenhagen
  - Klinikum St. Georg GmbH, Leipzig
  - Klinikum Leverkusen, Leverkusen
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Marburg, Marburg
  - Praxis Dr. med. Jens Taggeselle, Markkleeberg
  - Internistisches Facharztzentrum, Memmingen
  - Herz-Gefäß-Zentrum Nymphenburg, München
  - Marienkrankenhaus Klinikum St. Elisabeth, Neuwied
  - Kardiologische Gemeinschaftspraxis, Nienburg
  - Kardiologie am Weißen Turm, Nuremberg
  - Praxis für Innere Medizin, Nuremberg
  - Klinikum Nürnberg Süd, Nuremberg
  - via medis Nierenzentrum Oldenburg MVZ, Oldenburg
  - Fachärztin für Allgemeinmedizin, Osnabrück
  - MVZ Birkenallee, Papenburg
  - Internistische Gemeinschaftspraxis, Passau
  - Cardiologicum Prina, Pirna
  - Praxis Dr. med. Christoph Axthelm & Kollegen, Pirna
  - Paracelsus-Harz-Klinik, Quedlinburg
  - KardioPrax Remscheid, Remscheid
  - Zentrum für Prävention und Rehabilitation, Siegen
  - Studienzentrum der Herzklinik Ulm GbR, Ulm
  - Internistische Praxis Vellmar, Vellmar
  - Schwarzwald-Baar-Klinikum, Villingen-Schwenningen
  - Gemeinschaftspraxis Drs. Grosskopf, Wallerfing
  - Kliniken Nordoberpfalz AG, Weiden
  - Praxis Dr. med. Jörg Brosche, Weinböhla
  - Kardiologische Praxis Dr. med. Ayham Al Zoebi, Wermsdorf
  - Ev. Krankenhaus Witten gGmbH, Witten
- Switzerland (3):
  - Kantonsspital Aarau AG, Aarau
  - Kantonsspital Baden AG, Baden
  - Klinik Hirslanden, Zurich

IPD SHARING:
Plan to Share IPD: No